CLINICAL TRIAL: NCT06797739
Title: Effect of Nutritional Counseling and Mediterranean Diet on Patients With Diverticular Disease Evaluated Using the DICA Endoscopic Classification
Brief Title: Effect of Nutritional Counseling and Mediterranean Diet on Patients With Diverticular Disease
Acronym: Nutri-DICA
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Regione del Veneto - AULSS n. 7 Pedemontana (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 18987/22
Record Dates: First submitted 2023-04-07; First posted 2025-01-28 (Actual); Last update posted 2025-01-28 (Actual); Status verified 2025-01

CONDITIONS: Diverticular Diseases
Keywords: DICA endoscopic score; Medi-LITE score; Symptomatic Uncomplicated Diverticular Disease (SUDD)
MeSH Terms: conditions — Diverticular Diseases | interventions — Diet

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Dietary counselling on Mediterranean Diet (Experimental): Patients will be asked to follow the Mediterranean Diet and to participate to an educational program
  Interventions: Other: Nutritional counselling; Other: Diet
- Mediterranean Diet (Experimental): Patients will be asked to follow Mediterranean Diet only
  Interventions: Other: Diet
- Controls (No Intervention): Patients maintain their current lifestyle and dietary habits.

INTERVENTIONS:
Other: Nutritional counselling — Patients will be asked to follow the Mediterranean Diet and to participate to an educational program.
  Arms: Dietary counselling on Mediterranean Diet
Other: Diet — Patients will be asked to follow Mediterranean Diet only
  Arms: Dietary counselling on Mediterranean Diet; Mediterranean Diet

SUMMARY:
Diverticular Disease (DD) is a frequent condition in Western populations and may be associated with complications including bleeding, perforation, acute diverticulitis, and colon strictures. Severity of diverticular disease and its association with prognosis in relation to surgery using the Diverticular Inflammation and Complication Assessment (DICA) classification has been validated in several studies. A sedentary lifestyle, poor fibre intake and other unhealthy dietary habits have been associated with DD. On the contrary, the Mediterranean Diet (MD), which involves factors such as consuming locally grown food products, family meals, conviviality, involvement in the preparation of meals, as well as high intake of vegetables, legumes, fruit and cereals, medium intake of fish, low intake of meat and saturated fat, high intake of unsaturated fat (particularly olive oil), a medium-low intake of dairy products (yogurt and cheese), and a moderate intake of wine, seems to protect against DD. Moreover, populations that follow the MD pattern show a 50% lower rate of cardiovascular mortality due to cardiovascular disease and show highest longevity. A common finding in clinical practice is that a majority of patients undergoing a new diet stop to correctly follow the diet in the long term, suggesting the importance of periodic counselling for patients.

The aim of the study is to evaluate the impact of MD on DD and on severity of DD, and to explore the impact of incorporating a dietitian-driven counselling program in this condition.

DETAILED DESCRIPTION:
The investigators will verify whether a 12-week nutritional intervention is able to reduce DD-related symptoms, improve patient's quality of life and reduce the need for medication. DD severity will be assessed using DICA, MD adherence will be assessed with Medi-Lite (Mediterranean Literature scoring system), symptoms will be assessed with a VAS (visual analogue scale) questionnaire and IBS-SSS (the irritable bowel syndrome severity scoring system), nutritional status will be evaluated using BIA (bioelectrical impedance analysis) and metabolic blood parameters.

ELIGIBILITY:
Inclusion Criteria:

* Have given written informed consent to participate
* Diagnosis of SUDD deﬁned as the presence of symptoms (mainly abdominal pain, but also constipation, diarrhea and bloating) in patients with a previous diagnosis of diverticular disease at colonoscopy in the absence of any current complications (stenoses, abscesses, ﬁstulas)
* DICA assessment during a colonoscopy

Exclusion Criteria:

* Acute or complicated diverticulitis
* Hospitalized patients
* Patients with active oncological diseases.
* Former partial or total colonic resection or other surgical procedures for DD
* Short bowel syndrome or active perianal fistulas
* Female patients who are pregnant or breastfeeding
* Patients with known malabsorption diseases (e.g. celiac disease)
* Any unstable or uncontrolled cardiovascular, pulmonary, hepatic, renal, gastrointestinal, genitourinary, hematological, coagulation, immunological, endocrine/metabolic, or other medical disorder that, in the opinion of the investigator, would confound the study results or compromise patient safety
* Any surgical procedure requiring general anesthesia within 30 days prior to enrollment or is planning to undergo major surgery during the study period
* Patients undergoing a specific diet (e.g. diet for diabetics)
* Patients with known and well-established food allergies or intolerance to dietary elements of MD
* Patients with recent diagnosis of or non-controlled lactose intolerance
* Active participation in other interventional or drug research projects in the study period.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2023-04-04 (Actual); Primary Completion 2024-12-16 (Actual); Study Completion 2025-04-04 (Estimated)

PRIMARY OUTCOMES:
Remission of symptoms | 12 weeks
  The percentage of patients that will achieve symptom-free remission of symptoms
Adherence to diet | 12 weeks
  The effect of a counselling program on Medi-LITE score
DICA and diet | 12 weeks
  The differences in response based on basal DICA (Diverticular Inflammation and Complication Assessment, value 1-3, with DICA 3 meaning a worse outcome).

SECONDARY OUTCOMES:
Inflammation | 12 weeks
  To determine the percentage of patients with a reduction of fecal calprotectin
Metabolism | 12 weeks
  The percentage of patients with a modification in blood metabolic parameters: liver and renal function, cholesterol, HDL, LDL, triglycerides, glucose, HOMA (homeostasis model assessment) index, albumin.
Drug use | 12 weeks
  The percentage of patients with modifications in drug therapy.

CONTACTS AND LOCATIONS:
Overall Officials: Antonio Ferronato, MD, Principal Investigator — UOSD Endoscopia - Ospedale Alto Vicentino - AULSS 7 Pedemontana
Locations (1):
- UOSD Endoscopia - Ospedale Alto Vicentino - AULSS 7 Pedemontana, Santorso, Vicenza, Italy

IPD SHARING:
Plan to Share IPD: No
Individual participant data must be submitted to local Ethical Committee

REFERENCES:
- [Background] Tursi A, Brandimarte G, Di Mario F, Lanas A, Scarpignato C, Bafutto M, Barbara G, Bassotti G, Binda GA, Biondi A, Biondo S, Cassieri C, Crucitti A, Dumitrascu DL, Elisei W, Escalante R, Herszenyi L, Kruis W, Kupcinskas J, Lahat A, Lecca PG, Maconi G, Malfertheiner P, Mazzari A, Mearin F, Milosavljevic T, Nardone G, Chavez De Oliveira E, Papa A, Papagrigoriadis S, Pera M, Persiani R, Picchio M, Regula J, Stimac D, Stollman N, Strate LL, Walker MM; DICA International Group. The DICA Endoscopic Classification for Diverticular Disease of the Colon Shows a Significant Interobserver Agreement among Community Endoscopists: an International Study. J Gastrointestin Liver Dis. 2019 Dec 19;28(suppl. 4):39-44. doi: 10.15403/jgld-558. PMID 31930224
- [Background] Tursi A, Brandimarte G, Di Mario F, Elisei W, Picchio M, Allegretta L, Annunziata ML, Bafutto M, Bassotti G, Bianco MA, Colucci R, Conigliaro R, Dumitrascu D, Escalante R, Ferrini L, Forti G, Franceschi M, Graziani MG, Lammert F, Latella G, Maconi G, Nardone G, Camara de Castro Oliveira L, Chaves Oliveira E, Papa A, Papagrigoriadis S, Pietrzak A, Pontone S, Poskus T, Pranzo G, Reichert MC, Rodino S, Regula J, Scaccianoce G, Scaldaferri F, Vassallo R, Zampaletta C, Zullo A, Piovani D, Bonovas S, Danese S; DICA International Group. Prognostic performance of the 'DICA' endoscopic classification and the 'CODA' score in predicting clinical outcomes of diverticular disease: an international, multicentre, prospective cohort study. Gut. 2022 Jul;71(7):1350-1358. doi: 10.1136/gutjnl-2021-325574. Epub 2021 Oct 26. PMID 34702716
- [Background] Sofi F, Dinu M, Pagliai G, Marcucci R, Casini A. Validation of a literature-based adherence score to Mediterranean diet: the MEDI-LITE score. Int J Food Sci Nutr. 2017 Sep;68(6):757-762. doi: 10.1080/09637486.2017.1287884. Epub 2017 Feb 9. PMID 28276908